CLINICAL TRIAL: NCT04951336
Title: Multicenter Double-Blind, Placebo-Controlled RCT of Fomitopsis Officinalis/Trametes Versicolor for COVID-19
Brief Title: RCT of Mushroom Based Natural Product to Enhance Immune Response to COVID-19 Vaccination
Acronym: MACH19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Gordon Saxe, Director, Krupp Center for Integrative Research, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 200633-1c
Record Dates: First submitted 2021-06-30; First posted 2021-07-06 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: COVID-19 Vaccination

STUDY DESIGN:
Intervention Model Description: Mix model involving two groups and multiple measurements across study time-points
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mushrooms (Experimental): Drug: FoTv The dosage of FoTv is 8 capsules three times a day for 4 consecutive days. It does not need to be consumed with food. It is best taken at least 30 minutes before OR at least 60 minutes after meals, in the morning, noon and evening. Accidentally missed doses will not need to be taken at a later time but will be recorded in a daily diary. Should swallowing capsules be an issue, they can be opened and dispensed into water or juice for easy ingestion.
  Interventions: Dietary Supplement: FoTv
- Placebo (Placebo Comparator): Placebo: organic brown rice The dosage of Placebo is 8 capsules three times a day for 4 consecutive days. It does not need to be consumed with food. It is best taken at least 30 minutes before OR at least 60 minutes after meals, in the morning, noon and evening. Accidentally missed doses will not need to be taken at a later time but will be recorded in a daily diary. Should swallowing capsules be an issue, they can be opened and dispensed into water or juice for easy ingestion.
  Interventions: Dietary Supplement: FoTv

INTERVENTIONS:
Dietary Supplement: FoTv — Fomitopsis Officinalis and Trametes Versicolor

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial to evaluate the effect of two polypore mushrooms, Fomitopsis officinalis and Trametes versicolor (FoTv), for use as an adjunct to vaccination for COVID-19 in a general population at the time of COVID-19 vaccination.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical trial to evaluate the effect of two polypore mushrooms, Fomitopsis officinalis and Trametes versicolor (FoTv), for use as an adjunct to vaccination for COVID-19 in a general population at the time of COVID-19 vaccination.

Fo and Tv have immunomodulatory properties which may increase antibody titers in response to vaccination more than vaccination alone. However, because they are also immunomodulatory - not purely immune-stimulating - they may have the added benefit of simultaneously decreasing vaccine-related side effects following COVID-19 vaccination.

The study aims to establish the safety and feasibility of the use of FoTv vs placebo; evaluate the effect on post-vaccination clinical symptoms and immune response in 45 total subjects.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for or planning on scheduling COVID-19 vaccination
* Age 18 years and older
* Willing to avoid alcohol, cannabis, and dairy products during the study product in-take period.
* Capable of documenting vitals, symptoms, and study product intake daily and communicating this information to the study team

Exclusion Criteria:

* Known liver disease (or diagnosis of cirrhosis)
* Known renal disease or acute nephritis.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shubov, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mushrooms | Placebo
Started | 52 | 38
Completed | 51 | 38
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mushrooms | Placebo | Total
Number analyzed (Participants) | 52 | 38 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (15.6) | 33.5 (13.9) | 39.03 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 21 | 52
  Male | 21 | 17 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 41 | 26 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 52 | 38 | 90
Aspartate Aminotransferase (AST) Normal [Number; unit: participants] — Normal: ≤ 40 U/L; Abnormal: > 40 U/L
  participants | 50 | 38 | 88
Alanine Transaminase (ALT) Normal [Count of Participants; unit: Participants] — Normal: ≤ 41 U/L; Abnormal: > 40 U/L
  Participants | 43 | 34 | 77
Alkaline Phosphatase (ALP) Normal [Count of Participants; unit: Participants] — Normal: ≤ 129 U/L; Abnormal: > 129 U/L
  Participants | 52 | 36 | 88
Adjusted glomerular filtration rate (Adj. eGFR) Normal [Count of Participants; unit: Participants] — Normal: > 60 mL/min; Abnormal: <= 60 mL/min
  Participants | 38 | 35 | 73

OUTCOME MEASURES:

1. Primary Outcome: AST Normal to Abnormal Transition
Description: The Normal to Abnormal percentage reflects the percentage of participants with normal values at Day 1 that transitioned to abnormal at Day 14 relative to all participants with normal values at baseline.
Time Frame: 14 days
Population: Number of participants who were normal at baseline. Participants who were abnormal at baseline were excluded, therefore the number of participants in this analysis is different from the total number of participants in the Mushrooms or Placebo groups described in the study arms/groups.
Measure: Number; unit: % of participants who transitioned
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 50 | 38
% of participants who transitioned | 2.0 | 2.6
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; ratio of frequencies = 0.04

2. Primary Outcome: ALT Normal to Abnormal Transition
Description: The Normal to Abnormal percentage reflects the percentage of participants with normal values at Day 1 that became abnormal at Day 14 relative to all participants with normal values at baseline.
Time Frame: 14 days
Population: Number of participants who were normal at baseline. Participants who were abnormal at baseline were excluded.
Measure: Number; unit: % of participants who transitioned
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 43 | 34
% of participants who transitioned | 4.7 | 5.9
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; ratio of frequencies = 0.06

3. Primary Outcome: ALP Normal to Abnormal Transition
Description: as for outcome 2
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: % of participants who transitioned
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 52 | 36
% of participants who transitioned | 1.9 | 0
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 1.000, Chi-squared, Corrected; ratio of frequencies = 0.70

4. Primary Outcome: eGFR Normal to Abnormal Transition
Description: as for outcome 2
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: % of participants who transitioned
Arm/Group | Mushrooms | Placebo
Number analyzed (Participants) | 38 | 35
% of participants who transitioned | 10.5 | 2.9
Statistical Analysis 1: Comparison: Mushrooms vs Placebo; Test type: Superiority; p = 0.359, Chi-squared, Corrected; ratio of frequencies = 1.68

5. Secondary Outcome: SARS-CoV-2 Receptor Binding Domain (RBD)
Description: higher scores indicate higher levels of RBD levels
Time Frame: Single-dose vaccine (J&J): days 1, 14, and 28, and 6-months post-vaccination; two-dose vaccine (Pfizer or Moderna): days 1, 14, and 42 (two weeks after second dose), and 6-months post-vaccination; and vaccine booster: days 1, 3, and 14, and 6-months.
Population: Five participants (3 in the Active group and 2 in the Placebo group) had 1 or more antibody test results that were considered outliers, and these participants were excluded from further antibody and side-effect analyses.
Measure: Mean (Standard Deviation); unit: binding antibody units/mL
Groups:
- Active-Exposed; Active-Unexposed: Participants were classified as either previously exposed (memory responses) or unexposed (primary responses) and analyzed within and across Exposure Strata. At baseline, participants with detectable anti-CoV-2 Abs were deemed "previously exposed" and those with no or very low anti-CoV-2 Abs "previously unexposed." Active received supplementation with FoTv.
- Placebo-Exposed; Placebo-Unexposed: Participants were classified as either previously exposed (memory responses) or unexposed (primary responses) and analyzed within and across Exposure Strata. At baseline, participants with detectable anti-CoV-2 Abs were deemed "previously exposed" and those with no or very low anti-CoV-2 Abs "previously unexposed." Placebo received supplementation with placebo (brown rice).
Arm/Group | Active-Exposed | Active-Unexposed | Placebo-Exposed | Placebo-Unexposed
Number analyzed (Participants) | 30 | 19 | 25 | 11
binding antibody units/mL
  Day1 | 355.02881 (358.066647) | 1.29801 (1.937670) | 206.22357 (188.893233) | 1.35671 (2.474966)
  Day3: number analyzed (Participants) | 14 | 0 | 13 | 0
  Day3 | 541.90950 (456.766094) |  | 289.80001 (217.354133) |
  Day14 | 10116.05971 (6190.370668) | 700.61000 (2530.473761) | 10052.95574 (4834.742085) | 168.23960 (161.993614)
  Day28: number analyzed (Participants) | 16 | 18 | 11 | 11
  Day28 | 9674.97316 (5860.432037) | 3953.50332 (3460.118026) | 10469.33030 (3844.263396) | 5129.00732 (5704.361365)
  6month: number analyzed (Participants) | 23 | 14 | 17 | 10
  6month | 3209.48933 (3720.168648) | 6178.44885 (8273.702523) | 3398.50612 (4093.456937) | 3359.28725 (5108.022295)
Statistical Analysis 1: Comparison: Active-Exposed vs Active-Unexposed vs Placebo-Exposed vs Placebo-Unexposed; The LME analysis compared antibodies between two grouping factors, (1) Treatment Group (FoTv vs. Placebo) and (2) Exposure Stratum (previously exposed vs. unexposed), across four time points (days 3, 14, 28, and 6 months). At baseline, participants with detectable anti-CoV-2 antibodies were deemed "previously exposed" and those with no or very low anti-CoV-2 Abs "previously unexposed." Accordingly, all longitudinal analyses excluded baseline antibody data; Test type: Superiority — age was included as a covariate; p = 0.002, Mixed Models Analysis — Differences were considered statistically significant for p-values <0.05; F(2,150)=6.374. The analysis was repeated using log-transformed values and the resultant p value was also < 0.05

6. Secondary Outcome: SARS-CoV-2 Spike Protein ("Spike").
Description: higher scores indicate higher levels of Spike levels
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: binding antibody units/mL
Arm/Group | Active-Exposed | Active-Unexposed | Placebo-Exposed | Placebo-Unexposed
Number analyzed (Participants) | 30 | 19 | 25 | 11
binding antibody units/mL
  Day1 | 247.56807 (258.452559) | 0.47756 (0.400992) | 149.40025 (119.995872) | 0.78453 (1.023236)
  Day3: number analyzed (Participants) | 14 | 0 | 13 | 0
  Day3 | 380.70020 (307.487759) |  | 205.36409 (143.342600) |
  Day14 | 4488.11297 (1542.141350) | 392.53283 (1047.729456) | 4877.87445 (1549.014480) | 224.88593 (242.109014)
  Day28: number analyzed (Participants) | 16 | 18 | 11 | 11
  Day28 | 3981.34227 (1366.702076) | 1958.70983 (1542.192284) | 4719.52003 (1192.604423) | 2383.29307 (2275.359574)
  6month: number analyzed (Participants) | 23 | 14 | 17 | 10
  6month | 1544.40689 (1341.873844) | 2107.24372 (2696.389743) | 1546.52328 (1347.920386) | 1400.07776 (1673.265928)
Statistical Analysis 1: Comparison: Active-Exposed vs Active-Unexposed vs Placebo-Exposed vs Placebo-Unexposed; LME analysis compared antibodies between two grouping factors, (1) Treatment Group (FoTv vs. Placebo) and (2) Exposure Stratum (previously exposed vs. unexposed), across four time points (days 3, 14, 28, and 6 months). At baseline, participants with detectable anti-CoV-2 antibodies were deemed "previously exposed" and those with no or very low anti-CoV-2 Abs "previously unexposed." Accordingly, all longitudinal analyses excluded baseline antibody data; Test type: Superiority — age was included as a covariate; p = 0.002, Mixed Models Analysis — p < 0.05; F(2,157)=4.286. The analysis was repeated using log-transformed values and the resultant p value was also < 0.05

7. Secondary Outcome: Side-Effect Number
Description: count of the number of CDC side effects associated with vaccine. higher scores indicate higher number of endorsed side effects. Count of: feeling feverish, low fever in the afternoon, alternating fever and chills, chills, fatigue, muscle aches, nausea, headaches, redness/swelling at injection site, and pain at injection site. The range was from zero to 10.
Time Frame: Days, 1, 2, 3, 4, 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active-Exposed | Active-Unexposed | Placebo-Exposed | Placebo-Unexposed
Number analyzed (Participants) | 30 | 19 | 25 | 11
units on a scale
  Day1 | 0.6333 (1.73172) | 0.2632 (0.56195) | 0.5200 (0.77028) | 0.4545 (0.52223)
  Day2 | 2.9333 (2.36254) | 1.4737 (1.4737) | 3.2000 (2.92973) | 1.2727 (2.68667)
  Day3 | 3.2000 (2.70886) | 2.0526 (2.14667) | 3.3200 (2.62552) | 4.5455 (3.20511)
  Day4 | 1.5000 (2.17747) | 1.0526 (1.71509) | 2.2000 (2.56580) | 1.9091 (1.70027)
  Day5 | 1.0333 (1.62912) | 0.0526 (0.22942) | 0.9200 (1.55242) | 0.6364 (0.67420)
Statistical Analysis 1: Comparison: Active-Exposed vs Active-Unexposed vs Placebo-Exposed vs Placebo-Unexposed; LME analysis compared symptoms between two grouping factors, (1) Treatment Group (FoTv vs. Placebo) and (2) Exposure Stratum (previously exposed vs. unexposed), across 5 time points (days 1-5); Test type: Superiority; p = 0.060, Mixed Models Analysis; F(8,325)=1.898. Age was included as a covariate in this analysis

8. Secondary Outcome: Side-Effect Severity
Description: Sum of the side effect severities for the CDC side effects associated with vaccine. higher scores indicate higher severity. The side effects included: feeling feverish, low fever in the afternoon, alternating fever and chills, chills, fatigue, muscle aches, nausea, headaches, redness/swelling at injection site, and pain at injection site. The scale for each side effect ranged from zero to 4. The total possible scale was zero to 40.
Time Frame: Days, 1, 2, 3, 4, 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active-Exposed | Active-Unexposed | Placebo-Exposed | Placebo-Unexposed
Number analyzed (Participants) | 30 | 19 | 25 | 11
units on a scale
  Day1 | 1.0333 (3.06800) | 0.2632 (0.56195) | 0.6800 (1.14455) | 0.4545 (0.52223)
  Day2 | 3.7600 (3.53883) | 2.4000 (5.34255) | 7.0000 (7.08520) | 4.0000 (7.12741)
  Day3 | 4.6667 (5.93257) | 2.0000 (4.01386) | 5.6400 (5.38424) | 8.3636 (8.88001)
  Day4 | 1.5667 (3.16972) | 0.7895 (1.43678) | 3.5600 (5.49303) | 2.5455 (2.84125)
  Day5 | 0.9333 (1.70057) | 0.0526 (0.22942) | 1.2400 (2.61852) | 0.9091 (1.22103)
Statistical Analysis 1: Comparison: Active-Exposed vs Active-Unexposed vs Placebo-Exposed vs Placebo-Unexposed; Test type: Superiority — LME analysis compared symptoms between two grouping factors, (1) Treatment Group (FoTv vs. Placebo) and (2) Exposure Stratum (previously exposed vs. unexposed), across 5 time points (days 1-5); p = 0.326, Mixed Models Analysis; F(8,309)=1.156. Age was included as a covariate in this analysis

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Mushrooms | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/38
Other Adverse Events (participants affected / at risk) | 8/52 | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mushrooms (N=52) | Placebo (N=38)
ER visit (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — ER visit
hospitalization (Reproductive system and breast disorders) | 0 (0) | 0 (0) — hospitalization
Urgent Care Visit (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — urgent care visit
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mushrooms (N=52) | Placebo (N=38)
ALP Normal to Abnormal Transition (Hepatobiliary disorders) | 1 (1) | 0/36 (0) — Transitioning from normal function at baseline to abnormal function at 14 days. ALP, alkaline phosphatase. Participants who were abnormal at baseline were excluded.
AST Normal to Abnormal Transition (Hepatobiliary disorders) | 1/50 (1) | 1 (1) — Transitioning from normal function at baseline to abnormal function at 14 days. AST, aspartate aminotransferase. Participants who were abnormal at baseline were excluded.
ALT Normal to Abnormal Transition (Hepatobiliary disorders) | 2/43 (2) | 2/34 (2) — Transitioning from normal function at baseline to abnormal function at 14 days. ALT, alanine transaminase. Participants who were abnormal at baseline were excluded.
eGFR Normal to Abnormal Transition (Renal and urinary disorders) | 4/38 (4) | 1/35 (1) — Transitioning from normal function at baseline to abnormal function at 14 days. eGFR, estimated glomerular filtration rate, based on 2021 criteria. Participants who were abnormal at baseline were excluded.

LIMITATIONS AND CAVEATS:
Because of the rapidly changing nature of the COVID-19 pandemic, we didn't have sufficient time to ascertain, and stratify randomization based on, exposure status. Earlier launch might also have resulted in a larger proportion of Unexposed participants in the total sample.

A 4-day treatment regimen was selected. Alternate dosing regimens at time of and immediately post-vaccination might have yielded different effects on Ab and other outcomes.

we didn't examine Ab levels beyond 6-months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT04951336/Prot_SAP_000.pdf